CLINICAL TRIAL: NCT00677768
Title: A Multicenter Study for the Validation of ALS Biomarkers
Brief Title: Validation of Biomarkers in Amyotrophic Lateral Sclerosis (ALS)
Acronym: BIO_ALS-01
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: ALS Association (Other); ALS Therapy Alliance (Other); National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, James D. Berry MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: BIO_ALS-01; 5RC1NS068179-02 (NIH)
Record Dates: First submitted 2008-05-09; First posted 2008-05-14 (Estimated); Last update posted 2016-06-03 (Estimated); Status verified 2016-06

CONDITIONS: Amyotrophic Lateral Sclerosis; Lou Gehrig's Disease; Primary Lateral Sclerosis; Nervous System Diseases; Hereditary Spastic Paraparesis
Keywords: Biomarkers; Plasma; Cerebrospinal Fluid; DNA; Serum
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease; Nervous System Diseases; Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 650 blood samples (plasma and serum)will be collected from four groups: ALS volunteers diagnosed with ALS, volunteers with pure lower or pure upper motor neuron diseases, volunteers with other neurological diseases and healthy control volunteers.
  300 cerebrospinal fluid (CSF) samples will be collected from all four groups: ALS volunteers diagnosed with ALS, volunteers with pure lower or pure upper motor neuron diseases, volunteers with other neurological diseases and healthy control volunteers.
  Up to 600 DNA samples will also be collected from all 4 groups: ALS volunteers diagnosed with ALS, volunteers with pure lower or pure upper motor neuron diseases, volunteers with other neurological diseases and healthy control volunteers.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Early ALS
  Interventions: Other: No intervention
- Suspected ALS
  Interventions: Other: No intervention
- Disease Mimics of ALS
  Interventions: Other: No intervention
- Healthy Controls
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Sample collection

SUMMARY:
The purpose of this study is to collect 650 blood and 300 cerebrospinal fluid (CSF) samples from people with amyotrophic lateral sclerosis (ALS), pure lower or upper motor neuron diseases, as well as other neurodegenerative diseases and from people with no neurological disorder. Through comparison of these samples, the researchers hope to learn more about the underlying cause of ALS, as well as find unique biological markers, which could be used to diagnose ALS and monitor disease progression.

Additionally, up to 600 blood samples will be collected for a sub-study for DNA analysis. Studying components of the blood, such as DNA, may help us understand what happens when genes function abnormally and how it might be related to disease.

DETAILED DESCRIPTION:
Researchers tested what changes happen in volunteers with ALS that can be seen in the blood and what changes are unique to ALS and are different from those found in healthy volunteers and volunteers with neurological diseases other than ALS. These changes are called biomarkers. Biomarkers for ALS have been found in blood collected in earlier phases of this study. Biomarkers are non-genetic elements in your blood that may help to make diagnosing ALS easier. In the next phase, comparison of these changes in the blood of volunteers with ALS and without ALS will be used to confirm these biomarkers and to develop a tool to diagnose and monitor progression of ALS.

ELIGIBILITY:
1. ALS Volunteers

   Inclusion Criteria:
   * Diagnosis of possible (excluding volunteers with UMN signs ONLY), probable, probable-laboratory supported, or definite ALS, either sporadic or familial according to revised El Escorial criteria
   * Disease duration of less than or equal to two years from symptom onset
   * Age 30-80 years at the time of disease onset
   * Ability to provide informed consent
   * Ability to comply with study procedures
   * Medically safe to have lumbar puncture (lumbar puncture volunteers only)

   Exclusion Criteria:
   * Clinical evidence of chronic liver or renal failure
   * Presence of a bleeding disorder, problems with CSF pressure, allergy to local anesthetics, or a topical or other skin infection at the LP site (lumbar puncture volunteers only)
   * Use of any anti-platelet or anticoagulant drugs, such as plavix, aggrenox, ticlid, warfarin or coumadin (lumbar puncture volunteers only)
2. Suspected ALS (PMND) Volunteers

   Inclusion Criteria:
   * Diagnosis of suspected ALS defined as presence of UMN or LMN signs alone and the diagnosis of Clinically Probably Laboratory-Supported ALS CANNOT be proven by evidence in clinical grounds in conjunction with electrodiagnostic, neurophysiologic, neuroimaging or clinically laboratory studies
   * Disease duration of less than or equal to four years from symptom onset
   * Age 30-80 years at time of disease onset
   * Ability to provide informed consent
   * Ability to comply with study procedures
   * Medically safe to have lumbar puncture (lumbar puncture volunteers only)

   Exclusion Criteria:
   * Clinical evidence of chronic liver or renal failure
   * Genetically confirmed diagnosis of hereditary spastic paraparesis or spinal motor atrophy (SMA) disease
   * Presence of a bleeding disorder, problems with CSF pressure, allergy to local anesthetics, or a topical or other skin infection at the LP site (lumbar puncture volunteers only)
   * Use of any anti-platelet or anticoagulant drugs, such as plavix, aggrenox, ticlid, warfarin or coumadin (lumbar puncture volunteers only)
3. Neurological Disease Mimic Volunteers

   Inclusion Criteria:

   Diagnosis of one of the following:

   Pure Lower Motor Neuron Disease (LMND) mimics:
   * Multi-focal motor neuropathy
   * Autoimmune motor neuropathy
   * Cervical or lumbosacral radiculopathies

   Peripheral mononeuropathies:
   * Ulnar neuropathy
   * Carpal tunnel syndrome/median neuropathy
   * Peroneal neuropathy
   * Sciatic neuropathy
   * Spinal muscular atrophy
   * Spinobulbar muscular atrophy (Kennedy's disease)
   * Charcot Marie-Tooth Disease (CMT)

   Pure Upper Motor Neuron Disease (UMND) mimics:
   * Cervical myelopathy
   * Multiple sclerosis
   * Hereditary spastic paraparesis
   * Age 30-80 years
   * Ability to provide informed consent
   * Ability to comply with study procedures
   * Medically safe to have lumbar puncture (lumbar puncture volunteers only)

   Exclusion Criteria:
   * Diagnosis of suspected, possible, probable or definite ALS either sporadic or familial
   * Presence of positive family history of ALS
   * Clinical evidence of chronic renal or liver failure
   * Presence of a bleeding disorder, problems with CSF pressure, allergy to local anesthetics, or a topical or other skin infection at the LP site (lumbar puncture volunteers only)
   * Use of any anti-platelet or anticoagulant drugs, such as plavix, aggrenox, ticlid, warfarin or coumadin (lumbar puncture volunteers only)
4. Healthy Control Volunteers Inclusion Criteria

   * Absence of a known neurological disorder.
   * Age 30 - 80 years.
   * Ability to provide informed consent.
   * Ability to comply with study procedures.
   * Medically safe to have lumbar puncture.

Exclusion Criteria:

* History of ALS, myopathy, neuropathy, ALS mimic disorder or other neurodegenerative disease.
* Presence of positive family history of ALS.
* Clinical evidence of chronic liver or renal failure.
* Presence of bleeding disorder, problems with CSF pressure, allergy to local anesthetics, or a topical or other skin infection at the LP site (LP research volunteers only).
* Research participant must not be taking anti-platelet or anticoagulant drugs, such as plavix, aggrenox, ticlid, warfarin or coumadin (LP research volunteers only).

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be invited to participate in this study by their neurologists either in clinic or at a regular scheduled appointment visit.
Sampling Method: Non-Probability Sample
Enrollment: 475 (Actual)
Dates: Start 2008-04; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
ALS Functional Rating Scale (ALSFRS-R) | Every 6 months
  The ALSFRS-R is a quickly administered (5 min) ordinal rating scale used to determine a subject's assessment of their capability and independence in 12 functional activities. There are 12 questions, graded by the subject 0-4 (4 is normal). Score of 0 (worst) to 48 (best). Reflects speech and swallowing, fine motor skills, large motor skills, and breathing.

CONTACTS AND LOCATIONS:
Overall Officials: James D. Berry, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (30):
- United States (29):
  - Phoenix Neurological Associates, Ltd., Phoenix, Arizona
  - University of California Irvine, Orange, California
  - Mayo Clinic Neurology, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Lahey Clinic, Burlington, Massachusetts
  - Saint Mary's Healthcare, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Saint Louis University, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Robert Wood Johnson/UMDNJ, New Brunswick, New Jersey
  - Upstate Clinical Research, LLC, Albany, New York
  - Beth Israel Medical Center, PACC, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Carolinas Health Care, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - OSU Medical Center, Columbus, Ohio
  - Providence ALS Clinic, Portland, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - Pennsylvania State University, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Methodist Neurological Institute, Houston, Texas
  - University of Utah, Salt Lake City, Utah
- Montreal Neurological Institute, Montreal, Quebec, Canada

REFERENCES:
- See also: ALS Association Website — http://www.alsa.org
- See also: NEALS ALS Consortium — http://www.alsconsortium.org/